CLINICAL TRIAL: NCT06291896
Title: A Multicentric, Prospective Clinical Investigation to Evaluate Microwave Imaging Via MammoWave® in a Population-based Screening Program for Early Breast Cancer Detection to Make Breast Cancer Screening More Accurate, Inclusive, and Female-friendly
Brief Title: A Clinical Investigation to Evaluate Microwave Imaging Via MammoWave® in a Population-based Screening Program for Early Breast Cancer Detection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umbria Bioengineering Technologies (Industry)
Collaborators: London South Bank University (Other); ELAROS 24/7 Limited (UK) (Unknown); Servicio De Salud De Castilla La Mancha (Spain) (Unknown); IMT School for Advanced Studies Lucca (Other); EVITA - Cancro Hereditário (Portugal) (Unknown); Fondazione Toscana Life Sciences (Italy) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UBT 2023-01
Record Dates: First submitted 2024-02-19; First posted 2024-03-04 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Women's Health: Neoplasm of Breast

STUDY DESIGN:
Intervention Model Description: Clinical Investigation with class IIa medical device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): All participants perform:
  conventional breast examination path (i.e., screening mammogram, integrated with other radiological/histological output when deemed necessary by the responsible Investigator in each site) AND MammoWave exam.
  Interventions: Device: MammoWave

INTERVENTIONS:
Device: MammoWave — Women undergoing conventional breast screening examination will be asked by the clinical staff if they are interested in taking part in the study.
  A short visit should be performed to check the inclusion/exclusion criteria, review demographic data, and the volunteer's medical history. After performing this visit, the volunteers will perform the MammoWave exam on both their breasts.
  The exam will be composed of two phases: data acquisition and data processing. During the acquisition, which should take about 8 minutes, the volunteers would be lying down in a prone position, on the bed which is part of MammoWave.
  When the acquisition is completed, the data will be processed through a dedicated microwave imaging algorithm. The output will be composed of microwave images, plus parameters describing the images. MammoWave output will also comprise a label obtained using an optimized classification algorithm.

SUMMARY:
This is an open, multicentric, interventional, prospective, non-randomized clinical investigation. The first aim of the study is to confirm that MammoWave reaches sensitivity>75% and specificity>90% in breast cancer (BC) detection on 10.000 volunteers undergoing regular screening programs.

DETAILED DESCRIPTION:
MammoWave is a non-CE marked device that uses low-power (1mW) microwaves (1-9 GHz) instead of ionizing radiation (X-ray) for BC screening. MammoWave uses safe low-power radio frequency signals in the microwave band; it is a Class IIa medical device (non-invasive device). The previous generation of MammoWave had obtained the CE mark; in this investigation, the device contains the same hardware and will be used with the same acquisition method as the CE marked device, but additional data processing software will be used.

The 10,000 volunteers undergoing conventional breast screening examination will also undergo the MammoWave exam. The MammoWave results (WSF: breast With Suspicious Finding,i.e. with suspicious lesion, or NSF: No Suspicious Finding, i.e. breast without lesion or with low suspicious lesion) will be checked against the Reference Standard, to be intended as the output of conventional breast examination path (i.e., screening mammogram, integrated with other radiological/histological output when deemed necessary by the responsible Investigator in each site). Reference Standard may be BC+ for the histology-confirmed breast cancer (BI-RADS 6); BC- otherwise (BI-RADS 1, 2, 3).

(NOTE: BIRADS 4 and 5 are only image suspicion criteria: when a biopsy is performed, BIRADS are transformed in 6 (BC+) or 1,2 and 3 (BC-))

This clinical trial is performed within MammoScreen project [1] awarded in the context of HORIZON-MISS-2021-CANCER-02-01. UBT Srl is a partner of a Consortium which comprises (in addition to UBT): Toscana Life Sciences Foundation (Italy); London South Bank University (UK); ELAROS 24/7 Limited (UK); Servicio De Salud De Castilla La Mancha (Spain); Scuola IMT Alti Studi Lucca (Italy); EVITA - Cancro Hereditário (Portugal).

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 45 and 74 years
* Asymptomatic
* Signed informed consent form before starting any study activity
* Average risk of BC (every woman except those with know BRCA1, 2, TP53, and/or previous BC)
* Mammographic test, either 2D FFDM or 3D Digital Breast Tomosynthesis (DBT) (collecting oblique mediolateral projection [MLO] of the right breast, craniocaudal projection [CC] of the right breast, MLO projection of the left breast, CC projection of the left breast), performed within the past month with available results or planned to be performed in the same day of the MammoWave test or in the subsequent days
* Spontaneous willingness to comply with CIP and recommendations

Exclusion Criteria:

* Woman with breast prostheses
* Women with symptoms or some sign of suspected BC
* Women with BRCA1, 2, TP53 or previous BC
* Pregnant women
* Women who do not have mammographic manifestation of the tumor (known occult breast tumor with only axillar manifestation)
* Women with breast size larger than the largest MammoWave cup size

Ages: 45 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
MammoWave® sensitivity | During the procedure
  MammoWave® sensitivity (percentage of 'true positive' results) while using an optimized classification algorithm. The Reference Standard is intended as the output of conventional breast examination path (i.e. screening mammogram, integrated with other radiological/histological output when deemed necessary by the responsible Investigator). Reference Standard may be: BC+ for the histology-confirmed and classified as BI-RADS 1,2 or 3.
MammoWave® specificity | During the procedure
  MammoWave® specificity (percentage of 'true negative' results) while using an optimized algorithm.

SECONDARY OUTCOMES:
Detection rates by type of lesion | During the baseline
  Evaluation of the detection rates (sensitivity) according to the type of radiological finding (microcalcification, mass, asymmetry or architectural distortion group), also by breast density (according to BI-RADS ACR classification assigned by the radiologist), and comparison with the other standard screening and diagnostic modalities.
Recall rate | During the baseline
  Evaluation of MammoWave recalls, also by breast density (according to BI-RADS ACR classification assigned by the radiologist), and comparison with the other standard screening and diagnostic modalities.
Positive-predictive value | During the baseline
  Evaluation of MammoWave positive predictive value (for the biopsies performed), also by breast density (according to BI-RADS ACR classification assigned by the radiologist), and comparison with the other standard screening and diagnostic modalities.
Program screening rate | During the baseline
  Program screening rate, calculated as the proportion of women diagnosed with BC in the study population
BC detection rates of each by histological type and size of the BC and BI-RADS classification, also by breast density | During the baseline
  BC detection rates of each by histological type and size of the BC and BI-RADS classification, also by breast density
MammoWave® sensitivity and specificity after retrospective AI adjustment using the data at the end of the study | During the baseline
  Evaluation of the improvement in both sensitivity and specificity when retrospectively using AI algorithms for the evaluation of MammoWave® data after its further optimization with all data collected in the participants included in the study.
Agreement between different evaluator (i.e. local versus central) | During the baseline
  Evaluation of the reproducibility of results comparing the lectures performed at the study centers and the centralized lectures
Volunteers' satisfaction questionnaire | During the baseline
  Volunteers' satisfaction through a properly designed questionnaire collecting women's issues and plus during the exam with MammoWave® in the language spoken by the women

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (2):
  - Ospedale San Giovanni Battista - USL Umbria 2, Foligno, Perugia
  - IRCCS Policlinico San Martino, Genova
- Pomeranian Medical University Hospital, Szczecin, Poland
- Portugal (2):
  - Champalimaud Foundation, Lisbon
  - Clínica Dr. Passos Ângelo in Lisbon, Lisbon
- Spain (3):
  - Hospital Universitario Reina Sofía- Córdoba, Córdoba
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Hospitalario Universitario de Toledo, Toledo
- Diagnostic and Interventional Radiology, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Alvarez Sanchez-Bayuela D, Fernandez Martin J, Tiberi G, Ghavami N, Giovanetti Gonzalez R, Cruz Hernanez LM, Aguilar Angulo PM, Martinez Gomez AD, Rodriguez Sanchez A, Bigotti A, Khalesi B, Pontoriero L, Calabrese M, Tagliafico AS, Romero Castellano C. Microwave imaging for breast cancer screening: protocol for an open, multicentric, interventional, prospective, non-randomised clinical investigation to evaluate cancer detection capabilities of MammoWave system on an asymptomatic population across multiple European countries. BMJ Open. 2024 Nov 2;14(11):e088431. doi: 10.1136/bmjopen-2024-088431. PMID 39488412
- See also: [1] — https://mammoscreenproject.eu/